CLINICAL TRIAL: NCT07349498
Title: Cardiovascular Outcomes and Risk Evaluation Among Recipients of Hematopoietic Stem Cell Transplantation (CORE-HCT): A Prospective Multicenter Observational Study
Brief Title: Cardiovascular Outcomes and Risk Evaluation Among Recipients of Hematopoietic Stem Cell Transplantation
Acronym: CORE-HCT
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Hematology Hospital of Chinese Academy of Medical Sciences (Hematology Research Center of Chinese Academy of Medical Sciences) (Unknown); First Affiliated Hospital of Zhejiang University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology (Unknown); Xinqiao hospital of the third military medical university (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); Sun Yat-sen University Cancer Center, Sun Yat-sen University (Unknown); Sichuan Provincial People's Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Chinese PLA General Hospital (Other); Peking University Shenzhen Hospital (Other); Peking University Third Hospital (Other); Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, MD, Peking University People's Hospital
Other Study IDs: 2025-z232
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic Stem Cell Transplantation; Transplant Complication; Cardiovascular Events

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing hematopoietic stem cell transplantation: Patients who undergo allogeneic hematopoietic stem cell transplantation at participating medical center.

SUMMARY:
This is a prospective, multicenter observational study for recipients of hematopoietic stem cell transplantation. Patients who underwent hematopoietic stem cell transplantation at the participating centers will be entrolled in the study. The clinical characteristics, laboratory profiles, management measures, and clinical outcomes such as post-transplant cardiovascular events will be prospectively collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo hematopoietic cell transplantation at any of the participating medical centers.

Exclusion Criteria:

* Any other conditions that, in the opinion of the investigator, can interfere with the interpretation of data.
* Patient request to withdraw from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergo hematopoietic cell transplantation at any of the participating medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2036-06-30 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | At 30 days, 100 days, 3 months, 6 months, 1 years, 3 years, 5 years post hematopoietic stem cell transplantation.
  Major adverse cardiovascular events (MACE) after hematopoietic stem cell transplantation.

SECONDARY OUTCOMES:
Cardiovascular events | At 30 days, 100 days, 3 months, 6 months, 1 years, 3 years, 5 years post hematopoietic stem cell transplantation.
  Cardiovascular events after hematopoietic stem cell transplantation, such as cardiovascular death, ischemic heart disease, coronary artery disease, stroke, heart failure, arrhythmia cardiomyopathy, myocarditis, endocarditis, valvular heart disease, and pericardial disease.
Overall survival | At 30 days, 100 days, 3 months, 6 months, 1 years, 3 years, 5 years post hematopoietic stem cell transplantation.
  Overall survival after hematopoietic stem cell transplantation.
Event-free survival | At 30 days, 100 days, 3 months, 6 months, 1 years, 3 years, 5 years post hematopoietic stem cell transplantation.
  Events were defined as the occurrence of any of the following after allo-HSCT: grade III-IV acute graft-versus-host disease (GVHD), chronic GVHD requiring systemic immunosuppression, relapse or progression of the hematologic disease, or death from any cause during follow-up.
Complications of hematopoietic stem cell transplantation | At 30 days, 100 days, 3 months, 6 months, 1 years, 3 years, 5 years post hematopoietic stem cell transplantation.
  Complications arising from hematopoietic stem cell transplantation range from early issues such as regimen toxicity and acute GVHD to late effects including chronic GVHD, organ dysfunction, and secondary malignancies.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Xinqiao hospital of the third military medical university, Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - First Affiliated Hospital Xi'an Jiaotong University, Xi'an, Shaanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Hematology Hospital of Chinese Academy of Medical Sciences (Hematology Research Center of Chinese Academy of Medical Sciences), Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided